CLINICAL TRIAL: NCT07224126
Title: Technology Assisted Treatment for Trichotillomania: Open Trial
Brief Title: Technology Assisted Treatment of Trichotillomania: Open Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HabitAware Inc. (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Kent State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1943; R44MH114773 (NIH)
Record Dates: First submitted 2025-10-31; First posted 2025-11-04 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Trichotillomania
Keywords: hair pulling disorder; BFRB; Body-Focused Repetitive Behavior; trichotillomania; trich
MeSH Terms: conditions — Trichotillomania; Trichomonas Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-Arm Intervention: Keen2 Predictive Awareness Bracelet (Experimental): Participants in this single-arm study will receive a Keen2 awareness bracelet and companion mobile app for an 8-week period. During the first 4 weeks, participants will use the device to detect hair-pulling episodes and record contextual details (such as time, emotional state, activity, and location) after each detection. In the second 4 weeks, participants will receive predictive vibration alerts generated from their prior behavioral patterns. These alerts are designed to prompt preventive actions across three domains: (1) stimulus control (reducing environmental triggers), (2) competing response training (engaging hands in alternative behaviors), and (3) coping strategies (using relaxation or cognitive techniques).
  Interventions: Behavioral: Keen2 Predictive Awareness Bracelet

INTERVENTIONS:
Behavioral: Keen2 Predictive Awareness Bracelet — The Keen2 is a wrist-worn awareness bracelet paired with a mobile app that helps individuals with trichotillomania recognize and reduce hair-pulling behavior. The bracelet uses motion sensors to detect hand movements consistent with pulling and delivers gentle vibration alerts to increase awareness. During the first four weeks, participants log contextual information about each detected episode, including emotional state, location, and activity. Based on these data, the system delivers predictive vibration alerts during weeks five through eight to prompt behavior change strategies across three domains: (1) stimulus control, (2) competing response training, and (3) coping strategies.

SUMMARY:
This open-label feasibility trial evaluates the use of the Keen2 awareness bracelet for adults with trichotillomania (hair-pulling disorder). Participants will use the bracelet for eight weeks. During the first four weeks, they will wear the device and log contextual information (such as emotions, location, and activity) after each detected hair-pulling episode. Based on these data, participants will then receive tailored predictive alerts designed to support use of stimulus control, competing responses, and coping strategies. The study will assess usability, adherence, and changes in self-reported hair-pulling severity and awareness.

DETAILED DESCRIPTION:
This single-arm study is designed to test the feasibility and preliminary behavioral impact of a digital awareness intervention for trichotillomania. Participants aged 18 and older who report recurrent hair-pulling will receive a Keen2 bracelet and companion mobile app for an eight-week period.

Phase 1 (Weeks 1-4): Participants will use the device to detect pulling episodes and will record contextual information (such as time of day, emotional state, and environmental triggers) in the app following each detection.

Phase 2 (Weeks 5-8): Using data from the first phase, the system will deliver individualized predictive vibration alerts when behavioral patterns suggest increased risk of pulling. Alerts correspond to three intervention domains: (1) Stimulus control (reducing environmental cues), (2) Competing response training (engaging hands in alternative actions), and (3) Coping strategies (implementing relaxation or cognitive techniques).

Primary outcomes include usability, adherence, and changes in hair-pulling severity measured by the Massachusetts General Hospital Hairpulling Scale (MGH-HPS) from baseline to week 8, with a follow up at week 12. Secondary outcomes include knowledge of interventional domains as well as qualitative feedback on device helpfulness.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age (criterion 1a) with a diagnosis of TTM (criterion 1b)
* Must reportEnglish as their primary language (criterion 2)
* Report no current pharmacological or psychosocial intervention targeting TTM symptoms OR a6-week course of either intervention modality without change in frequency,intensity, or dosage (criterion 3)
* Reliable and consistent access to the internet and/or mobile device permitting the participant to meet withsomeone virtually for 90 min.
* Must report owning/access to a mobilephone running on Apple's operating system (iOS)
* Identifies a support person that is able to be contacted is an emergency arises.
* Agrees to allow the Kent State research team to share home address, mobile number, andalternate number/email with HabitAware, Inc., for purposes of mailing Keen2device and setting up Keen2 system.

Exclusion Criteria:

* Current suicidal/homicidal ideation, intent, or plan
* a diagnosis of another psychiatric condition that may impeded a participant's ability to fully utilize the app (e.g., psychotic disorder, major depressive disorder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-01-09 (Estimated); Study Completion 2026-01-09 (Estimated)

PRIMARY OUTCOMES:
Change in Trichotillomania Symptom Severity (NIMH-TSS) | Baseline, Week 4, and Week 8
  The primary outcome is the change in total score on the NIMH Trichotillomania Symptom Severity Scale (NIMH-TSS) from baseline to week 8. The NIMH-TSS is a clinician-rated scale assessing the frequency, intensity, and distress associated with hair-pulling behavior. Higher scores indicate greater symptom severity. A reduction in score reflects improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychological Sciences, Kent, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to KSU page describing the study — https://www.ksuparc.org/habit-aware